CLINICAL TRIAL: NCT06154876
Title: Effect Of Cough Assist Device On Hemodynamic Status And Oxygen Saturation For Ventilated Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nour Reda Abdelmonem Hafez, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC./012/003526
Record Dates: First submitted 2023-11-15; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Pneumonia Childhood; Intensive Care Unit; Children

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cough assist device and designed chest physical therapy (Experimental): Cough assist device involved 3-5 cycles with insufflation/exsufflation pressure beginning with +15 cm H2O to -15 cm H2O and maximum pressure of +40 cm H2O to -40 cm H2O for 4-5 sets for pediatric patients .and percussion, vibration, end expiratory pressure and bed mobility exercise.
  Interventions: Device: Cough assist device
- Designed chest physical therapy (Active Comparator): Percussion, vibration, end expiratory pressure and bed mobility exercise.
  Interventions: Device: Cough assist device

INTERVENTIONS:
Device: Cough assist device — Cough assist device Cough Assist clears secretions from the lungs by gradually applying positive air pressure to the airway and then rapidly shifting to negative air pressure . The resulting high expiratory flow simulates a deep, natural cough.
  Designed chest physical therapy Percussion, vibration, end expiratory pressure and bed mobility exercise.
  Other Names: Designed chest physical therapy

SUMMARY:
Statement of the problem:

•Is there an effect of the cough assist device on Hemodynamic status and oxygen saturation for ventilated children? Null hypothesis There will be no effect of cough assist device on hemodynamic status and oxygen saturation for ventilated children.

DETAILED DESCRIPTION:
Subjects:

The study targets the children from both sexes.diagnosed with pneumonia in intensive care unit. Sample size estimation will be carried out to determine the recruited number of children, selected randomly from Cairo University pediatric specialized hospital, Cairo to participate in the study.

Study design:

Randomized controlled clinical trial. Children will receive intervention type randomly,25 child will receive traditional chest physical therapy (postural drainage, percussion and vibration, end expiratory pressure) and bed mobility exercise.and the other 25 child will receive cough assist device in addition to traditional chest physical therapy (postural drainage, percussion and vibration, end expiratory pressure) and bed mobility exercise.

Children will be assessed by measuring heart rate, respiratory rate, blood pressure which reflect the physiological status, oxygen saturation,expired Tidal Volume and dynamic lung compliance which reflect clinical improvement of chest condition before and after receiving intervention

ELIGIBILITY:
Inclusion Criteria:

1. Children of both sexes, with age ranged from 4-9 years old.
2. Children will diagnosed with pneumonia.
3. Children will intubated on mechanical ventilation.
4. All children should be vitally stable during the study period.

Exclusion criteria:

Exclusion Criteria:

1. Hemodynamically unstable child.
2. Child with diaphragmatic hernia.
3. Child with pneumothorax (if chest tube is present).
4. Child with raised intracranial pressure.
5. Child with recent upper Gastrointestinal surgery

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Assessment of oxygen saturation | 14 days for each participant or time of weaning
  Pulse oximeter attached to the child and recorded oxygen saturation before and after intervention.
Assessment of expired Tidal Volume | 14 days for each participant or time of weaning
  Expired Tidal volume recorded from mechanical ventilation attached to the child before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nour Reda, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt